CLINICAL TRIAL: NCT02317835
Title: An Innovative System for the Early Identification, Monitoring, Evaluation and Diagnosis of Diabetic Foot Ulcers
Brief Title: Diabetic Foot Ulcer Prevention System
Acronym: DFUPS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: National Physical Laboratory (Other); University of South Wales (Other); Freeman Health System (Other); Pennine Acute Hospitals NHS Trust (Other); National Institute for Health Research, United Kingdom (Other Government); Photometrix (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: version 2 (02/3/2015)
Record Dates: First submitted 2014-12-10; First posted 2014-12-17 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot

ARMS (1):
- Study in healthy volunteers (Other): Skin foot temperature measurement by DFUPS device
  Interventions: Device: DFUPS

INTERVENTIONS:
Device: DFUPS — The DFUPS device is a two-camera instrument for capturing images of feet

SUMMARY:
To evaluate a recently developed non-invasive infrared thermal camera called Diabetic Foot Ulcer Prevention System (DFUPS) in a clinical setting by studying healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Has no history of diabetes
3. Has no previous history of foot ulceration
4. Has no previous history of foot surgery
5. Has palpable foot pulses on both feet (palpable posterior tibial artery pulse OR dorsalis pedis artery pulse OR both)
6. Has no history of peripheral neuropathy
7. Has no history of peripheral arterial disease
8. Must be able to provide meaningful written informed consent for the study

Exclusion Criteria:

1. Has active foot ulceration and infection
2. Has foot deformity which in the opinion of the Investigator, would interfere with interpreting the results of the study
3. Has any uncontrolled illness that, in the opinion of the Investigator, would interfere with interpreting the results of the study
4. Has an implantable electronic device
5. Is aged <18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-07; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Detection of hot spots on a foot thermal map image | 9 months

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - King's College Hospital, London
  - The Pennine Acute Hospitals NHS Trust, Manchester
  - The Newcastle upon Tyne Hospitals, Newcastle upon Tyne

REFERENCES:
- [Derived] Petrova NL, Whittam A, MacDonald A, Ainarkar S, Donaldson AN, Bevans J, Allen J, Plassmann P, Kluwe B, Ring F, Rogers L, Simpson R, Machin G, Edmonds ME. Reliability of a novel thermal imaging system for temperature assessment of healthy feet. J Foot Ankle Res. 2018 May 30;11:22. doi: 10.1186/s13047-018-0266-1. eCollection 2018. PMID 29854007